CLINICAL TRIAL: NCT05246254
Title: The Association of Preoperative Frailty Index and Incidence of Postoperative Delirium in Elderly Patients With Hip Fracture: a Prospective Cohort Study
Brief Title: Association of Frailty and Delirium in Elderly Hip Fracture Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Sponsor
Other Study IDs: BTCH-MZ-007
Record Dates: First submitted 2022-01-12; First posted 2022-02-18 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-02

CONDITIONS: Delirium in Old Age; Frailty
Keywords: frailty; postoperative delirium; hip fracture; elderly
MeSH Terms: conditions — Frailty; Emergence Delirium; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prefrailty group: According to the frailty index(FI) and FI =0.12~0.25
  Interventions: Diagnostic Test: Frailty index scale
- Frailty group: According to the frailty index(FI) and FI≥ 0.25
  Interventions: Diagnostic Test: Frailty index scale
- Nonfrailty group: According to the frailty index(FI) and FI<0.12
  Interventions: Diagnostic Test: Frailty index scale

INTERVENTIONS:
Diagnostic Test: Frailty index scale — There are clinically common scales for assessing weakness and delirium.
  Other Names: CAM scale; Nu-DESC sclae

SUMMARY:
Several studies have shown that frailty can be used as a marker for risk of adverse outcomes in elderly patients such as falls, disability, hospitalization, mortality, and can be used to predict patient clinical outcomes. The purpose of this study is to determine whether preoperative frailty can be used as a diagnostic and predictive factor for postoperative delirium in elderly patients with hip fracture.

DETAILED DESCRIPTION:
Frailty index (FI) is a reliable method to determine the assessment of frailty in elderly patients. Multiple prospective cohort studies have shown that frailty can be used as a marker for risk of adverse outcomes in older adults such as falls, disability, hospitalization, and mortality, and can be used to predict patient clinical outcomes. Whether frailty could be used as a diagnostic and predictive factor for delirium is urgently needed in a large population.

Therefore, this project intends to conduct a prospective cohort study. Patients will be divided into three groups according to frailty index (FI) before surgery, and delirium status will be evaluated by using scales after surgery, so as to explore the diagnostic and predictive value of frailty on POD. Once confirmed, the results of this study will be helpful for the early identification, screening, diagnosis and evaluation of treatment effect of POD. It is of great scientific significance and social benefit to reduce the incidence of POD, improve the prognosis of vulnerable patients and reduce the burden of disease.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were patients with hip fracture;
* Older than 65 years;
* Patients signed informed consent;
* American Society of Anesthesiologist (ASA) Rated I- III;
* The surgery was performed by the same anesthesia and surgical team.

Exclusion Criteria:

* Patients cannot sign the consent form or refuse to participate;
* A history of cognitive impairment;
* Unable to complete the cognitive function test;
* Mental disorder during initial assessment;
* Patients suffering from mental illness or substance use disorder;
* Incomplete or lost data during follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65 who underwent surgery for hip fractures
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium（POD） in elderly patients with hip fracture | Postoperative 7 days
  The percentage of the study population who developed delirium within seven days of surgery,postoperative delirium（POD） is defined according to the CAM criterion

SECONDARY OUTCOMES:
Duration of delirium | Postoperative 7 days
  The time between the first appearance of delirium
Delirium drug use | Postoperative 7 days
  dosage and name of medication prescribed by a neurologist
Length of hospital stay (HLOS) | Postoperative 30 days
  Collection of clinical data in the medical record
Length of ICU stay | Postoperative 30 days
  Collection of clinical data in the medical record
Hospital cost | Postoperative 30 days
  Expenses during hospitalization
Dindo-Clavien Classification{References:Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg 2004; 240(2):205-213.} | Postoperative 30 days
  Incidence of serious adverse reactions within 30 days after operation （the therapy used to correct a specific complication is the basis of this classification in order to rank a complication in an objective and reproducible manner.
  It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  Complications that have the potential for long-lasting disability after patient's discharge are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life.）
Death before and 30 days after discharge | 30 days after discharge
  Collection of clinical data in the medical record and follow-up update through telephone

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhang, PhD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided